CLINICAL TRIAL: NCT03820076
Title: Double Blind, Three Cohort, Placebo-controlled Trial to Assess Safety, Tolerance and Induced Bacterial Colony Counts of Three Ascending Doses of AZT-04 in Healthy Adult Volunteers
Brief Title: Safety Study of AZT-04 for Cosmetic Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azitra Inc. (Industry)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AZT04-001
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Study of Three Doses of AZT-04 for Skin Appearance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dose 1 (Experimental): AZT-04
  Interventions: Other: AZT-04
- dose 2 (Experimental): AZT-04
  Interventions: Other: AZT-04
- dose 3 (Experimental): AZT-04
  Interventions: Other: AZT-04

INTERVENTIONS:
Other: AZT-04 — Staphylococcus epidermidis

SUMMARY:
Double Blind, Three Cohort, Placebo-controlled Trial to Assess Safety, Tolerance and Induced Bacterial Colony Counts of Three Ascending Doses of AZT-04 in Healthy Adult Volunteers

DETAILED DESCRIPTION:
This is a single-center, prospective, double-blind, three cohort pilot study to assess the tolerability and induced changes in skin microbiome population and diversity of three ascending doses of test article code AZT-04 in normal, healthy subjects.

The study will consist of up to 7 scheduled study visits. There will be three cohorts in this study, each cohort composed of 6 subjects (total number of subjects is at least 18). Each cohort will be treated with both a placebo ointment and an ointment containing different concentrations of the Staphylococcus epidermidis. Approximately 1 ml of placebo ointment and 1 ml of AZT-04 ointment (test product composed of a commensal strain of Staphylococcus epidermidis) will be applied topically to two separate skin sites on the back, each site approximately 8 x 5 cm. Skin microbiome sampling will be performed before application of any test article (i.e., baseline) and each subsequent day for four (4) consecutive days. Samples will be shipped to a laboratory chosen by the Sponsor for analyses

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English, willing and able to read, understand, and sign the informed consent form
* Ability to complete the course of the study and comply with instructions
* Makes and Females ages 18-65 years, inclusively, in good general health as deemed by the investigator
* Individuals with Fitzpatrick skin type I, II, III, IV
* Individuals free of any systemic or dermatological disorder including a known history of allergies or other medical conditions which, in the opinion of the investigator, could interfere with the conduct of the study, interpretation of results or increase the risk of adverse reactions.
* Females practicing an acceptable method of birth control

Exclusion Criteria:

* individuals with any visible skin disease, skin condition including baseline erythema assessment > 0.5, or tattoos in the test area
* individuals with abnormal skin pigmentation at the test sites, which might interfere with subsequent evaluations of dermal responsiveness
* individuals with recent prolonged sun or tanning bed exposure in the test area
* individuals with excessive dryness or redness at the sites of application
* individuals with a known hypersensitivity to cosmetic or personal care formulations
* subjects must not have applied any lotions creams, powders, or oils to their backs the morning of the study. Additionally 2 hours must have passed since bathing or showering
* women who are pregnant or nursing
* individuals who have participated on a s study involving the test sites (back) in the previous 14 days
* individuals participating in another clinical study
* individuals with open or healing cuts/incisions abrasions, lesions, pustules, fissures or broken mucosa/skin in the test site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerance: mean erythema | 9 days
  to demonstrate the tolerability of three different doses of AZT-04 containing Staphylococcus epidermidis compared to placebo in healthy adult population--as s measured by mean erythema scores

SECONDARY OUTCOMES:
Bacterial Count | 9 days
  to assess the colonization of the test articles and placebo treated sites as it relates to the number of colony forming units (CFU's) over time after application and overall change in the microbiome diversity

CONTACTS AND LOCATIONS:
Locations (1):
- RCTS, Inc., Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided